CLINICAL TRIAL: NCT01693042
Title: Randomized Controlled Trial to Compare the Effects of Single Versus Repeated Intracoronary Application of Autologous Bone Marrow-derived Mononuclear Cells on Total and SHFM-predicted Mortality in Patients With Chronic Post-infarction Heart Failure
Brief Title: Compare the Effects of Single Versus Repeated Intracoronary Application of Autologous Bone Marrow-derived Mononuclear Cells on Mortality in Patients With Chronic Post-infarction Heart Failure
Acronym: REPEAT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, A. M. Zeiher, Prof. Dr. Andreas M. Zeiher, Johann Wolfgang Goethe University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-01-01REPEAT; 2011-000595-33 (EudraCT Number)
Record Dates: First submitted 2012-09-19; First posted 2012-09-26 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Heart Failure
Keywords: heart failure; old myocardial infarction; bone marrow-derived mononuclear cells; chronic; ischemic
MeSH Terms: conditions — Heart Failure; Bronchiolitis Obliterans Syndrome; Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single intracoronary cell application (Active Comparator): Single intracoronary application of autologous bone marrow derived mononuclear cells
  Interventions: Biological: intracoronary infusion of autologous bone marrow-derived cells
- repeated (2 times) intracoronary cell application (Active Comparator): 2 times (interval 4 months) intracoronary application of autologous bone marrow derived mononuclear cells
  Interventions: Biological: intracoronary infusion of autologous bone marrow-derived cells

INTERVENTIONS:
Biological: intracoronary infusion of autologous bone marrow-derived cells — Intracoronary infusion into open vessel / bypass supplying previous (> 3 months) infarct area
  Other Names: t2c001

SUMMARY:
Single or repeated application of autologous bone marrow-derived stem cells to treat chronic post-infarction heart failure

DETAILED DESCRIPTION:
Improve mortality and morbidity in patients with symptomatic chronic post-infarction heart failure under full dose conventional medical and device treatment including resynchronization therapy, by single versus repeated intracoronary infusion of autologous bone marrow-derived mononuclear cells.

ELIGIBILITY:
Inclusion Criteria:

* Previous myocardial infarction at least 3 months ago, open infarct vessel or bypass
* Left ventricular ejection fraction (LVEF) ≤ 45% on echocardiography
* Stable chronic heart failure NYHA class II to III under constant (4 weeks) evidence-based optimal medical treatment
* age 18 - 80 years
* written informed consent
* women of childbearing age: negative pregnancy test; effective contraception for the first 8 months in the trial

Exclusion Criteria:

* Non-ischemic cardiomyopathy
* Necessity for revascularization in other vessel than the infarct vessel at the time of study therapy
* Hemodynamic relevant severe valvular disease with indication for operative / interventional revision
* Heart failure with preserved ejection fraction (diastolic heart failure), LVEF > 45%
* Unstable Angina
* Severe peripheral artery occlusive disease (≥ Fontaine stadium III)
* Active infection (C-reactive protein > 10 mg/dl), chronic active hepatitis; any chronic inflammatory disease, HIV infection
* Neoplastic disease without documented remission in the last 5 years
* Stroke ≤ 3 months
* Impaired renal function (Serum creatinine > 2,5 mg/dl) at the time of study inclusion
* Relevant liver disease (GOT > 2x upper normal limit, spontaneous INR > 1,5).
* Diseases of hematopoetic system, anemia (Hemoglobin < 8.5 mg/dl), thrombocytopenia < 100.000/µl)
* Splenomegaly
* Allergy or intolerance of clopidogrel, prasugrel, ticagrelor, heparin, bivalirudin
* History of bleeding disorder
* gastrointestinal bleeding ≤ 3 months
* major surgery or trauma ≤ 3 months
* Uncontrolled hypertension
* Pregnancy, lactation period
* mental retardation
* previous cardiac cell therapy within last 12 months
* Participation in another clinical trial ≤ 30 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-11; Primary Completion 2022-11 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Mortality at 2 years after inclusion into the study | 2 years
  2-year observed mortality is significantly lower in patients receiving 2 repeated intracoronary applications of autologous bone marrow-derived cells (t2c001) compared to patients receiving 1 intracoronary application of autologous bone marrow-derived cells (t2c001)

SECONDARY OUTCOMES:
Morbidity at 2 and 5 years after inclusion into the study | 2 years and 5 years
  Efficacy endpoints:
  Comparison between the 2 treatment groups at 2-year and 5-year follow-up
  * Cardiac mortality, cardiovascular mortality
  * Rehospitalisation for heart failure
  * Ischemic cardiac events (STEMI, NSTEMI, ACS)
  * Coronary revascularisations (PCI / CABG)
  * Heart transplantation, Assist-device implantation
  * New resynchronization therapy, ICD implantation
  * NYHA-Status, NT-proBNP serum levels
  * Minnesota Living with Heart Failure Questionnaire
  Safety endpoints:
  bleeding events, all in-hospital events (during hospitalization for BMC therapy), life-threatening arrhythmias, new malignancies

CONTACTS AND LOCATIONS:
Overall Officials: Andreas M Zeiher, MD, Principal Investigator — Cardiology, Goethe University Frankfurt; Birgit Assmus, MD, Study Director — Cardiology, Goethe University Frankfurt
Locations (6):
- Germany (6):
  - Zentralklinik Bad Berka, Bad Berka
  - Goethe University Frankfurt, Frankfurt
  - Klinikum Fulda, Fulda
  - Universitätsklinikum Mainz, Mainz
  - Krankenhaus Hetzelstift, Neustadt
  - Zentralklinikum Suhl, Suhl